CLINICAL TRIAL: NCT04842591
Title: Characteristics of Pulmonary Vascular Changes in Patients With Kidney Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Other Study IDs: 33-022 ex 20/21
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension; Kidney Transplantation; Haemodialysis
Keywords: pulmonary hypertension; kidney transplantation; vascular remodeling; echocardiography; pulmo-renal axis
MeSH Terms: conditions — Hypertension, Pulmonary; Vascular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- kidney transplant candidates: Patients listed for first kidney transplantation
  Interventions: Diagnostic Test: exercise echocardiography

INTERVENTIONS:
Diagnostic Test: exercise echocardiography — All patients will undergo exercise echocardiography during a symptom-limited cardiopulmonary exercise test.

SUMMARY:
The aim of the study is to investigate pulmonary hemodynamics at rest and during exercise in patients before and after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* patients listed for first kidney transplantation at the Clinical Division of Nephrology

Exclusion Criteria:

* Age < 18 years
* combined organ transplantations (heart-kidney, pancreas-kidney etc.)
* patients with prior kidney transplantation
* high calcium score on cardiac-CT (> 160 Agatston Score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for kidney transplantation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the systolic pulmonary arterial pressure/cardiac output (SPAP/CO) slope | Baseline and 1 year after kidney transplantation
  Change in the systolic pulmonary arterial pressure/cardiac output (SPAP/CO) slope (calculated as the difference of maximal and resting SPAP divided by the difference of maximal and resting CO) before versus one year after kidney transplantation assessed by exercise echocardiography

SECONDARY OUTCOMES:
Change in systolic pulmonary arterial pressure at rest before versus one year after kidney transplantation assessed by (exercise) echocardiography | Baseline and 1 year after kidney transplantation
Change in systolic pulmonary arterial pressure at 25 Watts before versus one year after kidney transplantation assessed by (exercise) echocardiography | Baseline and 1 year after kidney transplantation
Change in mean pulmonary arterial pressure at rest before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in mean pulmonary arterial pressure during exercise before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in pulmonary vascular resistance at rest before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in pulmonary vascular resistance during exercise before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in pulmonary arterial wedge pressure at rest before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in pulmonary arterial wedge pressure during exercise before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in cardiac output at rest before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation
Change in cardiac output during exercise before versus one year after kidney transplantation | Baseline and 1 year after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Kovacs, MD, PhD, Principal Investigator — Medical University of Graz, Department of Internal Medicine, Division of Pulmonology
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Division of Pulmonology, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Background] Levey AS, Atkins R, Coresh J, Cohen EP, Collins AJ, Eckardt KU, Nahas ME, Jaber BL, Jadoul M, Levin A, Powe NR, Rossert J, Wheeler DC, Lameire N, Eknoyan G. Chronic kidney disease as a global public health problem: approaches and initiatives - a position statement from Kidney Disease Improving Global Outcomes. Kidney Int. 2007 Aug;72(3):247-59. doi: 10.1038/sj.ki.5002343. Epub 2007 Jun 13. PMID 17568785
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Clinical epidemiology of cardiovascular disease in chronic renal disease. Am J Kidney Dis. 1998 Nov;32(5 Suppl 3):S112-9. doi: 10.1053/ajkd.1998.v32.pm9820470. No abstract available.
- [Background] Wen CP, Cheng TY, Tsai MK, Chang YC, Chan HT, Tsai SP, Chiang PH, Hsu CC, Sung PK, Hsu YH, Wen SF. All-cause mortality attributable to chronic kidney disease: a prospective cohort study based on 462 293 adults in Taiwan. Lancet. 2008 Jun 28;371(9631):2173-82. doi: 10.1016/S0140-6736(08)60952-6. PMID 18586172
- [Background] O'Leary JM, Assad TR, Xu M, Birdwell KA, Farber-Eger E, Wells QS, Hemnes AR, Brittain EL. Pulmonary hypertension in patients with chronic kidney disease: invasive hemodynamic etiology and outcomes. Pulm Circ. 2017 Jul-Sep;7(3):674-683. doi: 10.1177/2045893217716108. Epub 2017 Jun 29. PMID 28660793
- [Background] Abassi Z, Nakhoul F, Khankin E, Reisner SA, Yigla M. Pulmonary hypertension in chronic dialysis patients with arteriovenous fistula: pathogenesis and therapeutic prospective. Curr Opin Nephrol Hypertens. 2006 Jul;15(4):353-60. doi: 10.1097/01.mnh.0000232874.27846.37. PMID 16775448
- [Background] Kawar B, Ellam T, Jackson C, Kiely DG. Pulmonary hypertension in renal disease: epidemiology, potential mechanisms and implications. Am J Nephrol. 2013;37(3):281-90. doi: 10.1159/000348804. Epub 2013 Mar 16. PMID 23548763
- [Background] Sise ME, Courtwright AM, Channick RN. Pulmonary hypertension in patients with chronic and end-stage kidney disease. Kidney Int. 2013 Oct;84(4):682-92. doi: 10.1038/ki.2013.186. Epub 2013 Jun 5. PMID 23739239
- [Background] Pabst S, Hammerstingl C, Hundt F, Gerhardt T, Grohe C, Nickenig G, Woitas R, Skowasch D. Pulmonary hypertension in patients with chronic kidney disease on dialysis and without dialysis: results of the PEPPER-study. PLoS One. 2012;7(4):e35310. doi: 10.1371/journal.pone.0035310. Epub 2012 Apr 18. PMID 22530005
- [Background] Abedini M, Sadeghi M, Naini AE, Atapour A, Golshahi J. Pulmonary hypertension among patients on dialysis and kidney transplant recipients. Ren Fail. 2013;35(4):560-5. doi: 10.3109/0886022X.2013.766567. Epub 2013 Feb 25. PMID 23438072
- [Background] Walther CP, Nambi V, Hanania NA, Navaneethan SD. Diagnosis and Management of Pulmonary Hypertension in Patients With CKD. Am J Kidney Dis. 2020 Jun;75(6):935-945. doi: 10.1053/j.ajkd.2019.12.005. Epub 2020 Mar 19. PMID 32199709
- [Background] Wolfe JD, Hickey GW, Althouse AD, Sharbaugh MS, Kliner DE, Mathier MA, Wu CM, Tevar AD, Soman P. Pulmonary vascular resistance determines mortality in end-stage renal disease patients with pulmonary hypertension. Clin Transplant. 2018 Jun;32(6):e13270. doi: 10.1111/ctr.13270. Epub 2018 May 15. PMID 29697854
- [Background] Foderaro AE, Baird GL, Bazargan-Lari A, Morrissey PE, Gohh RY, Poppas A, Klinger JR, Ventetuolo CE. Echocardiographic Pulmonary Hypertension Predicts Post-transplantation Renal Allograft Failure. Transplant Proc. 2017 Jul-Aug;49(6):1256-1261. doi: 10.1016/j.transproceed.2017.01.085. PMID 28735990
- [Background] Zlotnick DM, Axelrod DA, Chobanian MC, Friedman S, Brown J, Catherwood E, Costa SP. Non-invasive detection of pulmonary hypertension prior to renal transplantation is a predictor of increased risk for early graft dysfunction. Nephrol Dial Transplant. 2010 Sep;25(9):3090-6. doi: 10.1093/ndt/gfq141. Epub 2010 Mar 17. PMID 20299337
- [Background] Tang M, Batty JA, Lin C, Fan X, Chan KE, Kalim S. Pulmonary Hypertension, Mortality, and Cardiovascular Disease in CKD and ESRD Patients: A Systematic Review and Meta-analysis. Am J Kidney Dis. 2018 Jul;72(1):75-83. doi: 10.1053/j.ajkd.2017.11.018. Epub 2018 Feb 9. PMID 29429751